CLINICAL TRIAL: NCT05637606
Title: HIgh Versus STAndard Blood Pressure Target in Hypertensive High-risk Patients: The HISTAP Randomized Clinical Trial.
Brief Title: HIgh Versus STAndard Blood Pressure Target in Hypertensive High-risk Patients Undergoing Major Abdominal Surgery
Acronym: HISTAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Humanitas Clinical and Research Center (Other)
Collaborators: Societa Italiana Anestesia Analgesia Rianimazione e Terapia Intensiva (Other)
Responsible Party: Principal Investigator, Antonio Messina, Principal Investigator, Humanitas Clinical and Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HISTAP TRIAL
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Blood Pressure; Complication,Postoperative; Intraoperative Hypotension
Keywords: Blood pressure; Intraoperative Hypotension; Postoperative complications; Postoperative mortality
MeSH Terms: conditions — Postoperative Complications | interventions — Ephedrine; Norepinephrine

STUDY DESIGN:
Intervention Model Description: The study will be a multicentric, randomized, non-blinded clinical trial. Eligible patients will be assigned in a 1:1 ratio to either a to control or treatment group. Randomization list will be created by a computer with the use of a permuted block design and embedded in the Electronic Case Report Form. Randomization will be performed using a 'block of 6" and stratified according to predefined baseline characteristics:
  1. Age ≥ 75 years
  2. Preoperative systolic pressure
     1. < 140 mmHg
     2. ≥ 140 mmHg
Who Masked: Outcomes Assessor
Masking Description: The trial intervention is not blinded for investigators, clinical staff, and patients, as blinding intraoperative MAP target is not feasible. The physicians of each center assessing all postoperative outcomes will be masked for the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MAP 80 (Experimental): Intervention group: intraoperative mean blood pressure target > 80 mmHg. Treatment of hypotension (defined as a mean blood pressure of below 80 mmHg) using intravenous bolus or continuous infusion of vasopressors, or fluids using a dedicated algorithm considering the pulse pressure or stroke volume variation and the mini fluid challenge to optimize mean blood pressure values.
  Interventions: Drug: Ephedrine; Drug: Norepinephrine; Drug: Etilefrine Hydrochloride bolus; Diagnostic Test: Use of pulse pressure and stroke volume variation (PPV and SVV); use of Mini Fluid Challenge (mini_FC)
- MAP 65 (Other): Control group: intraoperative mean blood pressure target > 65 mmHg. Treatment of hypotension (defined as a mean blood pressure of below 65 mmHg) using intravenous bolus or continuous infusion of vasopressors, or fluids using a dedicated algorithm considering the pulse pressure or stroke volume variation and the mini fluid challenge to optimize mean blood pressure values.
  Interventions: Drug: Ephedrine; Drug: Norepinephrine; Drug: Etilefrine Hydrochloride bolus; Diagnostic Test: Use of pulse pressure and stroke volume variation (PPV and SVV); use of Mini Fluid Challenge (mini_FC)

INTERVENTIONS:
Drug: Ephedrine — In both the group, the target MAP can be maintained by means of bolus of ephedrine (2.5 mg). The maximal dose for the ephedrine allowed is 25 mg (10 boluses of 2.5 mg), after this threshold a continuous infusion of norepinephrine will be started
  Other Names: Ephedrine bolus
Drug: Norepinephrine — In both the group, the target MAP can be maintained by means of bolus of ephedrine (2.5 mg) or Etilefrine (1 mg). The continuous infusion of norepinephrine, as decided by the attending anesthetist, may be started at any point of the intraoperative period. The starting dose of norepinephrine is the lowest needed to reach the predefined MAP target.
  Other Names: norepinephrine infusion
Drug: Etilefrine Hydrochloride bolus — The maximal dose for the etilefrine allowed is 10 mg (10 boluses of 1 mg), after this threshold a continuous infusion of norepinephrine will be started
Diagnostic Test: Use of pulse pressure and stroke volume variation (PPV and SVV); use of Mini Fluid Challenge (mini_FC) — PPV, SVV and mini_FC will guide fluid bolus administration during an episode of intraoperative hypotension, following two predefined algorithms for laparotomic/non laparotomic surgery
  Other Names: Hemodynamic optimization

SUMMARY:
This study is a multicenter randomized controlled trial comparing two strategies of mean arterial blood pressure management (MAP ≥ 80mmHg vs MAP ≥ 65 mmHg) in high-risk surgical patients undergoing elective laparotomic/laparoscopic surgery.

DETAILED DESCRIPTION:
Intraoperative hypotension has been associated with major postoperative complications after non-cardiac surgery. However, is is still unclear the optimal intraoperative mean arterial pressure (MAP) target in the subgroup of those patient with an history of hypertension at home, and at risk of developing postoperative complications.

The objective of this study is to assess the effects of an intraoperative blood pressure management strategy aiming at keeping the MAP ≥ 80mmHg), as compared to the conventional practice (to maintain intraoperative MAP ≥ 65mmHg), on a composite outcome considering the death rate and the incidence of major events in patient scheduled for elective laparotomic/laparoscopic surgery.

The primary outcome is a composite of 30-days from operation mortality rate and at least one major organ dysfunction including the renal, respiratory, cardiovascular and neurologic systems or new onset of sepsis and septic shock occurring by day 7 after surgery.

ELIGIBILITY:
Inclusion criteria (all the following)

1. Adult patients ≥ 60 years
2. History of chronic hypertension requiring home therapy.
3. Scheduled for major elective abdominal surgery (laparoscopic, robotic or laparotomic)
4. Expected surgical duration of at least 3 hours.
5. Needing invasive arterial and hemodynamic monitoring as decided by the attending anesthetist, according to the rules of good clinical practice of each involved center.

AND

At increased risk of postoperative complications (at least one of the following):

1. American Society of Anesthesiologists (ASA) class 3 or 4
2. Known or documented history of coronary artery disease (angina, myocardial infarction or acute coronary syndrome).
3. Known or documented history of peripheral vascular disease.
4. Known or documented history of heart failure requiring treatment.
5. Ejection fraction less than 30% (echocardiography)
6. Signs of diastolic moderate to severe dysfunction or chronic hypertensive cardiomyopathy (echocardiography)
7. Moderate or severe valvular heart disease (echocardiography)
8. Diagnosis of Chronic Obstructive Pulmonary Disease (COPD) Radiographically confirmed or according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria.
9. Diabetes currently treated with an oral hypoglycemic agent and/or insulin
10. Morbid obesity (BMI ≥35 kg/m2)
11. Preoperative serum albumin <30 g/l
12. Anaerobic threshold (if done) <14 ml/kg/min
13. Exercise tolerance equivalent to six metabolic equivalents (METs) or less as defined by American College of Cardiology/American Heart Association guidelines

Exclusion criteria

1. Refusal of consent
2. Chronic kidney disease with glomerular filtration rate <30 ml/min/1.73 m2 or requiring renal-replacement therapy for end-stage renal disease
3. Acute cardiovascular event, including acute or decompensated heart failure and acute coronary syndrome (within prior 30 days).
4. Urgent or time-critical surgery
5. Aortic or Renal vascular surgery (including nephrectomy)
6. Liver Surgery
7. Neurosurgery
8. Surgery for palliative treatment only or ASA physical status 5
9. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of postoperative mortality and at least one major organ dysfunction (see description in the secondary outcomes). | up to 30 days after operation
  Composite postoperative outcome

SECONDARY OUTCOMES:
Hospital stay (days) | up to 30 days after operation
  Hospital stay (days)
ICU stay (days) | up to 30 days after operation
  Intensive Care Unit stay (days)
ICU readmission | up to 30 days after operation
  Intensive Care Unit readmissions
Sequential Organ Failure Assessment (SOFA) scores on postoperative | up to 7 days after operation
  Postoperative organ failure - SOFA scores ranges from 0 (<2% of mortality) to 24 (>90% of mortality)
Overall intraoperative fluid balance | day 1 after the operation
  Intraoperative infusions (crystalloids, colloids, blood products) / Intraoperative loss balance (urine output)
Mortality | up to 30 days after operation
  Mortality
Vasopressors use | day 1 after the operation
  Dose and timing of vasoactive drug infusion intraoperatively
Need for reoperation | day 30 after operation
  Need of a new surgical treatment

OTHER OUTCOMES:
CARDIOVASCULAR complications | day 7 after operation
  * Acute heart failure
  * Myocardial injury after non-cardiac surgery
  * Myocardial infarction
  * Bradycardia
  * Symptomatic proximal deep venous thrombosis
  * Peripheral arterial and venous thrombosis
NEUROLOGICAL complications | day 7 after operation
  * Stroke
  * Subarachnoid hemorrhage
  * Cerebral venous thrombosis
  * Seizure
  * Acute delirium
RESPIRATORY | day 7 after operation
  * Acute respiratory distress
  * Hypoxemia with or without acute respiratory distress
  * Need for invasive, non-invasive ventilation or high-flow nasal cannula for acute respiratory distress.
  * Acute respiratory distress syndrome.
  * Pulmonary edema
  * Pulmonary embolism
RENAL | day 7 after operation
  • Acute Kidney Injury (AKI) and AKI stages defined according to the AKIN classification/staging system of acute kidney injury
SEPSIS and Septic shock | day 7 after operation
  Based on the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3) criteria, sepsis required a quick Sequential Organ Failure Assessment (qSOFA) Score ≥ 2 points due to infection, septic shock defined as indicated by the Surviving Sepsis Campaign Guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Messina, Principal Investigator — Department of Biomedical Sciences, Humanitas University, Pieve Emanuele, Milano, Italy
Locations (18):
- Italy (18):
  - Ospedali Riuniti Foggia- Università di Foggia, Foggia, Apulia
  - Department of Anesthesia and Intensive Care, University Hospital of Modena, Modena, Emilia-Romagna
  - Policlinico A. Gemelli, Rome, Lazio
  - Humanitas Research Hospital, Rozzano, MILANO
  - Fondazione Istituto San Raffaele G. Giglio, Cefalù, Sicily
  - Careggi University Hospital, Florence, Tuscany
  - Unit of Anesthesiology and Intensive Care B, Department of Surgery, Dentistry, Gynecology and Pediatrics, AOUI-University Hospital Integrated Trust of Verona, Verona, Veneto
  - Azienda Ospedaliero - Universitaria SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Istituto Nazionale dei Tumori, Milan
  - Ospedale Antonio Cardarelli, Napoli
  - Azienda sanitaria Friuli Occidentale (AsFO], Pordenone
  - Ospedale Santo Stefano, Prato
  - Ospedale S. Anna di Castelnovo ne' Monti, Reggio Emilia
  - Sant'Eugenio ASL Roma 2:, Roma
  - Azienda Ospedaliero Universitaria di Sassari, Sassari
  - Ospedale Molinette, Torino
  - Ospedale Santa Chiara di Trento, Trento

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Messina A, Robba C, Calabro L, Zambelli D, Iannuzzi F, Molinari E, Scarano S, Battaglini D, Baggiani M, De Mattei G, Saderi L, Sotgiu G, Pelosi P, Cecconi M. Association between perioperative fluid administration and postoperative outcomes: a 20-year systematic review and a meta-analysis of randomized goal-directed trials in major visceral/noncardiac surgery. Crit Care. 2021 Feb 1;25(1):43. doi: 10.1186/s13054-021-03464-1. PMID 33522953
- [Background] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589